CLINICAL TRIAL: NCT06103851
Title: Investigation of the Effect of Mask Use on Temporomandibular Joint Functionality
Brief Title: Effect of Mask Use on Jaw Functionality
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, assist. prof., Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-4611
Record Dates: First submitted 2021-10-05; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Mask wearing; Temporomandibular joint disorder; TMJ; EMG
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to COVID-19 pandemic the use of masks has been made mandatory to prevent contagion. Individuals concluded that the use of masks has a negative effect on temporomandibular joint functions. In our literature search, we did not find any study on this subject. The aim of our study is to investigate the effect of mask use on temporomandibular joint function. Female individuals between the ages of 18-45 will be included in the research. Before participating in the study, individuals will be informed about the study and informed consent will be obtained.

Evaluations will be made twice a day, in the morning without the use of a mask, in the morning when using a mask, and in the evening (with the use of a mask for 6 hours, approximately 6 hours after the first assessment). Each individual to be measured will use the same brand and size N95 mask to be provided by us.

Evaluations: Individuals' m. masseter muscle activity with surface EMG, pain intensity felt in the jaw area, the pain threshold on m. masseter and m.temporalis will be evaluated. The questionnaire created by investigators also will be helded.

DETAILED DESCRIPTION:
The COVID-19 pandemic was declared by the World Health Organization (WHO) in March 2019. Due to the pandemic, the use of masks has been made mandatory to prevent contagion. We think that the use of masks has a negative effect on temporomandibular joint functions. In our literature search, we did not find any study on this subject. The aim of our study is to investigate the effect of mask use on temporomandibular joint function.

Female individuals between the ages of 18-45 working at Istanbul Medipol University will be included in the research. Before participating in the study, individuals will be informed about the study and informed consent will be obtained.

Evaluations will be made twice a day, in the morning without the use of a mask, in the morning when using a mask, and in the evening (with the use of a mask for 6 hours, approximately 6 hours after the first assessment). Each individual to be measured will use the same brand and size N95 mask to be provided by us.

Evaluations: Individuals' m. masseter muscle activity with surface EMG, pain intensity felt in the jaw area, the pain threshold on m. masseter and m.temporalis will be evaluated. The questionnaire created by investigators also will be helded.

Evaluation of Muscle Activity: M. masseter muscle activity will be recorded using the sEMG feature of the VitalStim device. Electrodes will be placed on the area where the muscle is swollen by maximizing the muscle contraction. The individual will be seated and rested for 5 minutes before sEMG recording and will be left for 1 minute without recording for the acclimatization period after electrode placement.

Pain Severity Assessment: the pain intensity of the participants will be questioned with a visual analog scale. On a ruler divided from 0 to 10 at equal intervals, the person will be asked to mark the degree of pain he feels in his jaw. According to the VAS, 0 means "no pain" and 10 means "as bad pain as possible".

Pressure Pain Threshold Assessment: Pressure pain threshold will be measured by the physiotherapist with a hand algometer (Baseline FDK 10) over M. Temporalis and M. Masseter. The algometer will be applied vertically to the most painful point, increasing the pressure by 1 kg/cm2 every three seconds until the patient feels pain, and the pressure value at which the pain begins will be recorded. 3 measurements will be made at 60 second intervals and the average value will be considered as the pain threshold.

Evaluation of Mandibular Opening: Maximum mandibular opening will be measured with the help of caliper at the final level of mouth opening, lateral deviation, protrusion and retrusion movements.

Self Designed Survey: A questionnaire consisting of open-ended, multiple-choice and likert-scale questions questioning the demographic information of individuals and the complaints/discomforts that may occur with the mask in the jaw joint will be administered via Google Forms, an online platform.

ELIGIBILITY:
Inclusion Criteria:

* who voluntarily agreed to participate in the study
* who is able to wear N95 mask for 6 hours

Exclusion Criteria:

* Those with chronic jaw pain
* Those who have had Covid-19 (due to ongoing joint pain)
* Acute jaw trauma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Among the academicians working in our institution, healthy participants aged between 18-45 and volunteering to participate in the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
surface EMG of masseter muscle | 6 weeks
  Masseter function with the VitalStim® Plus Electrotherapy System, the sEMG biofeedback activity of electrical impulses generated during the voluntary muscle contraction and relaxation cycle will be measured.
Pain intensity | 6 weeks
  Pain on jaw region that felt after face mask usage Individuals' pain intensity will be evaluated using a numerical analog scale ranging from 0 to none at all and 10 to very severe pain.

SECONDARY OUTCOMES:
pressure pain threshold | 6 weeks
  to the most painful point on masseter and temporalis muscle, algometer applied vertically, increasing the pressure by 1 kg/cm2 every three seconds until the patient feels pain, and the pressure value at which the pain begins will be recorded.
Jaw discomfort by face mask questionnaire | 6 weeks
  questionaire that collect demographic information of individuals and the complaints/discomforts that may occur with the mask usage around the jaw joint
maximum mouth opening | 6 weeks
  Individual opens the mouth as much as possible and the distance between front teeth are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Özdemir Görgü, PhD, Study Chair — Medipol University
Locations (1):
- Gizem Ergezen, Istanbul, Beykoz, Turkey (Türkiye)